CLINICAL TRIAL: NCT06396338
Title: Voluntary Surgical Terminations of Pregnancy: Comparison of the Hemorrhagic Risk Depending on the Term, Between 10 and 14 Weeks of Amenorrhea or Between 14 and 16 Weeks of Amenorrhea
Brief Title: Voluntary Surgical Terminations of Pregnancy: Comparison of the Hemorrhagic Risk Depending on the Term
Acronym: HEMOVG
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0167
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Voluntary Termination of Pregnancy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patient treated at the Toulouse University Hospital for an abortion: Patient treated at the Toulouse University Hospital for an abortion between 10 and 16 weeks (dating by ultrasound) presenting with a single and evolving pregnancy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire is offered to patients who meet the eligibility criteria and who have given their non-objection during the abortion request consultation.
  This questionnaire includes questions for screening for anxiety and depressive disorders.

SUMMARY:
Voluntary termination of pregnancy (abortion) is a major current societal issue. This is a very common situation, around 225,000 abortions are carried out every year in France. The legislation has recently been amended, with the law of March 2, 2022 aimed at strengthening the right to abortion (no. 2022-295) which extended the legal period for voluntary termination of pregnancy from 14 to 16 weeks amenorrhea (AS).

The National College of French Obstetrician Gynecologists (CNGOF), in a press release published on October 12, 2020 in response to the proposed law adopted by the National Assembly, wishes to draw attention to the fact that the procedure of surgical abortion between 14 and 16 AS changes nature. He states that additional procedures are necessary beyond 14 weeks, which could be a source of complications. In addition, the practice recommendations have not been updated following this extension of time, the centers performing abortions are therefore free regarding the protocol for carrying out these so-called late abortions (between 14 and 16 weeks).

There are two pregnancy termination techniques practiced in France: medical or surgical.

Due to the recent nature of these late abortions, practitioners still have little experience of the consequences of these procedures and this compromises the quality of the information provided to patients. It is necessary to have quality studies to improve knowledge about late-term abortions, in order to be able to correctly inform patients and allow them to make an informed choice regarding the method used.

This study follows the modification of the legislation extending the legal period for abortion, with the aim of providing arguments regarding the safety of carrying out surgical abortions at these more advanced stages of pregnancy.

In addition, abortion often generates anxiety, the term at which it is carried out could influence the experience of patients. This study would therefore also improve knowledge about the experience of abortion, in order to better support patients throughout their journey.

ELIGIBILITY:
Inclusion Criteria:

* Woman treated for the performance of a surgical abortion between 10 and 16 weeks (dating by ultrasound)
* Singleton pregnancy

Exclusion Criteria:

* Protected adult patient (guardianship, curatorship, safeguard of justice)
* Refusal to participate expressed by the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient coming at hospital for voluntary termination of pregnancy (abortion)
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of anxiety or depressive disorder | 3 weeks after abortion
  Anxiety will be measured using State-Trait Anxiety Inventory (STAI) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lola LOUSSERT-CHAMBRE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No